CLINICAL TRIAL: NCT03965780
Title: The Scleroderma Patient-centered Intervention Network - Scleroderma Support Group Leader EDucation Program Trial (SPIN-SSLED)
Brief Title: The SPIN - Scleroderma Support Group Leader EDucation Program Trial (SPIN-SSLED)
Acronym: SPIN-SSLED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Davis Institute (Other)
Responsible Party: Principal Investigator, Brett D Thombs, Professor, Faculty of Medicine, McGill University; Senior Investigator, Lady Davis Institute for Medical Research, Jewish General Hospital, Lady Davis Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-112A
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Scleroderma, Systemic
Keywords: Scleroderma; Systemic Sclerosis; Peer Support Group; Training
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental): Participants in the training group will receive a 13-week training program delivered via videoconference. The program includes 13 modules delivered via videoconference over the course of the 3-month program in weekly 60- to 90-minute sessions. Participants will receive a training manual, be shown filmed vignettes, and will have access to a chatroom and an online resource centre.
  Interventions: Other: SPIN-SSLED Program
- Wait-list control group (No Intervention): Participants in the wait-list control group will not receive the training program and will have no access to the resources indicated above.

INTERVENTIONS:
Other: SPIN-SSLED Program — The SPIN-SSLED Program is a 3-month-long (13 sessions) group training program designed to be delivered via videoconferencing to provide information and skills to improve leader support group leaders' confidence and self-efficacy to carry out their leadership roles and reduce the burden on them of leading a support group. Each session is about 90 minutes long and covers one of the 13 modules of the program.
  Module topics includes: (1) The Leader's Role; (2) Starting a Support Group; (3) Structuring a Support Group Meeting; (4) Scleroderma 101; (5) Successful Support Group Culture; (6) Managing Support Group Dynamics; (7) Loss and Grief: The support group leader; (8) Loss and Grief in Scleroderma: Supporting group members; (9) Advertising and Recruitment for the Support Group; (10) The Continuity of the Group; (11) Supporting Yourself as a Leader; (12) Remote Support Groups; and (13) Transitions in Support Groups.
  Other Names: Scleroderma Patient-centered Intervention Network - Scleroderma Support group Leader EDucation (SPIN-SSLED) Program
  Arms: Training group

SUMMARY:
Many people living with scleroderma, a rare autoimmune connective tissue disease, attend support groups to help them cope with the disease. Support groups provide a safe environment where people facing a similar challenge can come together to share disease-related experiences and exchange practical and emotional support. This is especially important for rare diseases such as scleroderma as organized support services can be limited.

However, many people with scleroderma do not have access to scleroderma support groups, and many support groups that are initiated are not sustained due to a number of obstacles. Leaders of these support groups play a particularly important role. They are responsible for a wide range of tasks including administrative details that go into planning meetings, facilitating effective and meaningful discussions, managing any issues that may arise in group dynamics, balancing their own needs with the needs of the group and many more.

The Scleroderma Patient-centered Intervention Network (SPIN) team has worked with patient organizations and an advisory team of scleroderma support group leaders to develop the Support group Leader EDucation (SPIN-SSLED) Program for scleroderma support group leaders with the goals of (1) providing information and resources to leaders to help them feel more comfortable, confident and supported in their roles and (2) to provide people with the skills they need to establish scleroderma support groups where none exist.

The SPIN-SSLED Trial will be used to evaluate the effectiveness of the SPIN-SSLED Program on scleroderma support group leaders' self-efficacy (primary outcome) in carrying out their leader tasks (which is defined as their perceived ability to carry out actions needed to be successful in support group leadership), burnout and emotional well-being.

DETAILED DESCRIPTION:
People with rare diseases face the same challenges as those with more common diseases plus unique challenges, including limited disease education and lack of specialized support options. Professionally organized support services for common diseases are often available through the healthcare system, but are not typically available in rare diseases. As a result, many people with rare diseases look to peer-led support groups for disease-specific education and support.

Support groups provide important benefits to people with burdensome medical conditions, based on the principle that people who face similar challenges can empower one another through emotional and practical support. Support groups may be held face-to-face or online, led by professionals or peers, and have a structured or an unstructured format. Activities typically involve an educational or information-sharing component and the exchange of emotional and practical support.

Systemic sclerosis (SSc), or scleroderma, is a rare, chronic, autoimmune connective tissue disease characterized by abnormal fibrotic processes and excessive collagen production. Peer-led support groups play an important role for many people with SSc. Currently, there are approximately over 250 leaders and co-leaders affiliated with SPIN-SSLED's partners Scleroderma Canada and Canadian provincial organizations, including Sclérodermie Québec, the Scleroderma Foundation (United States), Scleroderma & Raynaud's UK (United Kingdom), Scleroderma Australia and Australian state organizations, and Scleroderma New Zealand, almost all led by people with SSc. Many people with SSc, however, cannot access support groups, and many initiated support groups are not sustained due to challenges that could be addressed via leader training. SPIN partner organizations are committed to improving support group quality and access by providing training to existing support group leaders and to new leaders to start groups in underserved areas and via the Internet.

The SPIN-SSLED Program was developed by a team of researchers with expertise in SSc, patient organization representatives, and a Patient Advisory Board comprised of current SSc support group leaders. The program content and design are based on results of SPIN's preliminary research on support groups in SSc and informed by instructional material for support group leaders SPIN identified via the internet and by consultations with support group leaders. The program uses a problem-based learning approach. Problem-based learning is a learner-centered approach that integrates theory and practice by providing the necessary knowledge and skills, presenting a complex, real-world problem, then working to identify an approach to solving the problem. To implement this, each module, or learning session, will introduce a topic and provide an overview of key information. Then, there will be a guided discussion among training group participants about possible approaches and solutions. The program includes 13 modules that will be delivered live via webinar over the course of the 3-month program. In addition to the live modules, SPIN-SSLED participants will receive a workbook that summarizes didactic material that is provided and will be shown filmed vignettes demonstrating effective group facilitation techniques and ways to respond to support group issues. SPIN-SSLED participants will also have access to an online resource center that includes a range of helpful tools for leaders including files of SSc related videos to show at meetings and an online forum for leaders to post questions, open only to leaders enrolled in the training program.

The aim of the SPIN-SSLED Trial is to assess the effectiveness of the SPIN-SSLED Program on scleroderma support group leaders' self-efficacy (primary outcome), which SPIN defined as their perceived ability to carry out actions needed to be successful in support group leadership, burnout and emotional well-being. Additionally, participants will be asked about their satisfaction with the program.

SPIN's partners from the Scleroderma Canada, including Sclérodermie Québec, Scleroderma Foundation, Scleroderma & Raynaud's UK, Scleroderma Association of New South Wales and Scleroderma New Zealand will contact group leaders to describe the SPIN-SSLED Full-Scale Trial and ascertain interest in participating. They will also provide SPIN-SSLED personnel with a list of their support group leaders. SPIN-SSLED personnel will then send email invitations with the consent form to all support group leaders on these lists. Following this, support group leaders will be contacted by phone within 24 hours to describe the study, review the consent form, and answer questions any question they may have. SPIN will enroll 180 SSc support group leaders to participate in the trial. 90 participants will be randomized to the waitlist control group and 90 to the training group. Three groups will run simultaneously per 3-month period for a total of 15 months.

Based on SPIN's previous experience with videoconferencing and consistent with previous trials of videoconference training, to maximize effective interaction and participation, 6 group leaders will be assigned to each training group. Training sessions will be delivered using the GoToMeeting® videoconferencing platform, a high-performance platform that has been used successfully for similar applications.

A survey will be administered to all participants before the trial. Participants randomized to either the training group or waitlist control group will also be administered a baseline, post-intervention and 3-months post-intervention surveys for outcome measures. The first survey will contain a demographics questionnaire designed for this study that includes basic demographic information, such as gender, age and employment status and disease-related variables, such as years since scleroderma diagnosis as well as their general availabilities to attend the 60-90 minute sessions. All questionnaires will be completed using the online surveying tool Qualtrics. Once the online survey data is collected, data will be exported to the statistics software program, International Business Machines Corporation Statistical Package for the Social Sciences (IBM SPSS).

ELIGIBILITY:
Inclusion Criteria:

* Be a current scleroderma support group leader or have been identified by our partner patient organizations as a new leader
* Be available to participate at times when sessions are scheduled
* Be able to use the internet to access the training program
* Be English or French-speaking

Exclusion Criteria:

* Having a co-leader enrolled in trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
Leader Self-Efficacy: Scleroderma Support Group Leader Self-efficacy Scale (SSGLSS) | 3-months post-randomization
  Leader self-efficacy will be evaluated using the Scleroderma Support Group Leader Self-efficacy Scale (SSGLSS) which was developed by the SPIN research team, including the members of the SPIN Support Group Advisory Team, to measure support group leader self-efficacy for performing leader tasks. The SSGLSS is a 32-item scale is scored on a 6-point Likert scale from 1 (strongly disagree) to 6 (strongly agree) with possible total scores from 32 to 192 and higher scores indicating greater self-efficacy. The primary outcome analysis will compare SSGLSS scores between the intervention and waitlist control groups using a generalized linear random effects model, adjusted for baseline SSGLSS scores.

SECONDARY OUTCOMES:
Leader Self-Efficacy: Scleroderma Support Group Leader Self-efficacy Scale (SSGLSS) | 6-months post-randomization
  Leader self-efficacy will be evaluated using the Scleroderma Support Group Leader Self-efficacy Scale (SSGLSS) which was developed by the SPIN research team, including the members of the SPIN Support Group Advisory Team, to measure support group leader self-efficacy for performing leader tasks. The SSGLSS is a 32-item scale is scored on a 6-point Likert scale from 1 (strongly disagree) to 6 (strongly agree) with possible total scores from 32 to 192 and higher scores indicating greater self-efficacy. The primary outcome analysis will compare SSGLSS scores between the intervention and waitlist control groups using a generalized linear random effects model, adjusted for baseline SSGLSS scores.
Burnout | 3-months post-randomization and 6-months post-randomization
  Leader burnout will be measured by the Oldenburg Burnout Inventory (OLBI), which assesses exhaustion and disengagement due to burnout and has been validated in diverse populations (16 items, 4-point scale from 1 = strongly disagree to 4 = strongly agree). The OLBI was initially designed for work-related burnout but has been adapted for numerous settings and in multiple countries and languages. The SPIN research team revised the wording of each OLBI item to reflect the support group environment rather than a work environment (e.g., "I find my work to be a positive challenge" was revised to "I find my role as a support group leader to be a positive challenge"). The OLBI has a two-factor structure (exhaustion and disengagement) with good measurement properties. Higher scores indicate higher levels of exhaustion and disengagement. Internal consistency reliability (Cronbach's alpha) in patients with SSc was 0.84 for exhaustion and 0.80 for disengagement.
Leader Satisfaction with Leading a Support Group | 3-months post-randomization and 6-months post-randomization
  Leader satisfaction with leading a support group will be measured using a modified version of the participation efficacy subscale of the Volunteer Satisfaction Index (VSI). The original version of the VSI was validated using a sample of volunteers (N = 327) and was found to be reliable and constructually valid. As several other studies have done previously, we have modified the wording of some of the items to reflect participants' volunteer role as support group leaders. The participation efficacy subscale asks respondents to indicate their level of satisfaction on 7 items using a 7-point Likert scale from 1 (very dissatisfied) to 7 (very satisfied).
Emotional Distress | 3-months post-randomization and 6-months post-randomization
  Emotional distress will be evaluated using the Patient Health Questionnaire-8 (PHQ-8) items which measure depressive symptoms over the last 2 weeks on a 4-point scale, ranging from 0 (not at all) to 3 (nearly every day). Higher scores indicate more depressive symptoms. The PHQ-8 performs equivalently to the PHQ-9, which has been shown to be a valid measure of depressive symptoms in patients with scleroderma.
Participant Satisfaction: SPIN-SSLED Program | 3-months post-randomization
  Participant satisfaction with the SPIN-SSLED Program will be evaluated with the Client Satisfaction Questionnaire-8 (CSQ-8), a standardized survey that is used to assess satisfaction with health services. Items are scored on a Likert scale from 1 (low satisfaction) to 4 (high satisfaction) with total scores ranging from 8 to 32 and higher scores indicating greater satisfaction with the program. This measure will only be administered to participants in the intervention arm.

CONTACTS AND LOCATIONS:
Overall Officials: Brett D Thombs, PhD, Principal Investigator — Lady Davis Institute for Medical Research, McGill University
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 12 months after the collection of the primary outcome
Access Criteria: Approval of proposed purpose for data access

REFERENCES:
- [Background] Thombs BD, Aguila K, Dyas L, Carrier ME, Fedoruk C, Horwood L, Canedo-Ayala M, Sauve M, Kwakkenbos L, Malcarne VL, El-Baalbaki G, Pelaez S, Connolly K, Hudson M, Platt RW; SPIN-SSLED Support Group Advisory Team. Protocol for a partially nested randomized controlled trial to evaluate the effectiveness of the Scleroderma Patient-centered Intervention Network Support Group Leader EDucation (SPIN-SSLED) Program. Trials. 2019 Dec 12;20(1):717. doi: 10.1186/s13063-019-3747-z. PMID 31831073
- [Derived] Thombs BD, Levis B, Carrier ME, Dyas L, Konrad V, Sauve M, Benedetti A; SPIN-SSLED Support Group Advisory Team. Association of support group leader experience with Scleroderma Patient-centered Intervention Network Support group Leader EDucation Program outcomes: Secondary analysis of a two-arm parallel partially nested randomized controlled trial. J Scleroderma Relat Disord. 2024 Sep 4;10(1):65-74. doi: 10.1177/23971983241272742. eCollection 2025 Feb. PMID 39552943
- [Derived] Thombs BD, Levis B, Carrier ME, Dyas L, Nordlund J, Tao L, Aguila K, Bourgeault A, Konrad V, Sauve M, Connolly K, Henry RS, Ostbo N, Levis AW, Kwakkenbos L, Malcarne VL, El-Baalbaki G, Hudson M, Wurz A, Culos-Reed SN, Platt RW, Benedetti A; SPIN-SSLED Support Group Leader Advisory Team. Effects of a support group leader education program jointly developed by health professionals and patients on peer leader self-efficacy among leaders of scleroderma support groups: a two-arm parallel partially nested randomised controlled trial. Orphanet J Rare Dis. 2022 Oct 28;17(1):396. doi: 10.1186/s13023-022-02552-x. PMID 36307891

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/80/NCT03965780/Prot_SAP_000.pdf